CLINICAL TRIAL: NCT00274586
Title: Tolerability of a Four Weeks Treatment With Aggrenox® Modified Release Capsules b.i.d, Compared to Reduced Dose During the First Two Weeks of Treatment in a Double-Blind, Randomized Controlled Parallel Group Comparison Trial Among Taiwanese Patients With Previous TIAs or Ischemic Stroke
Brief Title: Headache Study to Compare Aggrenox Full Dose and Reduced Dose
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9.155
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Cerebrovascular Accident
MeSH Terms: conditions — Stroke

INTERVENTIONS:
Drug: Aggrenox® modified release capsules
Drug: Aggrenox® modified release capsules matching placebo

SUMMARY:
Tolerability of a four weeks treatment with Aggrenox® modified release capsules b.i.d, compared to reduced dose during the first two weeks of treatment in a double-blind, randomized controlled parallel group comparison trial among Taiwanese patients with previous TIA's or ischemic stroke.To monitor frequency and intensity of headaches and other safety parameters among Taiwanese patients with previous TIA's or ischemic stroke given Aggrenox using a titration scheme or not

DETAILED DESCRIPTION:
The major objective of the study is to evaluate the tolerance of headache and safety in Taiwan Taiwanese patients who are receiving two different dosing regimens of Aggrenox and Aggrenox placebo. The first group will start with placebo on days 1-4, daily dose on days 5-14, and following by b.i.d treatment on 15-28 days. This group will also receive a matching placebo in the morning and one Aggrenox capsule in the evening before on days 5-14. It enables to reduce the perception of dipyridamole-associated headache. The second group will receive the placebo twice daily on days 1-4, and medication twice daily for the remaining course. The third group will receive the placebo twice daily for the whole course.

Study Hypothesis:

NULL AND ALTERNATIVE HYPOTHESES

From a subject diary, asking for the most frequent side effects observed in the ESPS2 trial, the cumulative headache (intensity x frequency) per day based on the first three days of treatment period defines the primary endpoint.

I: H0: Median cumulative headache is equal for all treatment groups vs. HA: Median cumulative headache is not equal for all treatment groups

II: H0: Median cumulative headache of low dose regimen?Median cumulative headache of regular dose vs. HA: Median cumulative headache of low dose regimen < Median cumulative headache of regular dose

Comparison(s):

Compare Aggrenox full dose, reduced dose and placebo

ELIGIBILITY:
Inclusion Criteria:

1. 20 years old or above.
2. History of TIA or completed ischemic stroke
3. Signed informed consent.
4. Patient with score < 2 on modified Rankin's Classification of Neurological Status.

Exclusion Criteria:

1. Patients with known or suspected prior intracranial haemorrhage or history of brain injury or brain tumor.
2. Disorders related to syncope, drop attacks, congenital vascular malformation, aneurysm, angioma, or epilepsy, psychiatric disorders.
3. Peptic ulcer or gastrointestinal bleeding within 6 months.
4. History of hypersensitivity or intolerance to study drugs or aspirin.
5. Experienced habitual headache (any form) within the past 3 months.
6. History of dysphasia, dysphagia, dementia, or unconsciousness.
7. Patients currently taking other medications known to cause headaches (e.g., nitrates).
8. Patients with deteriorating angina, subvalvular aortic stenosis or hemodynamic liability (e.g., in conjunction with a recent myocardial infarction).
9. Uncontrolled hypertension (SBP > 220 mmHg, DBP> 120 mmHg) or life-threatening disease.
10. Any significant disorders, such as chronic renal failure (serum creatinine > 2.0 mg/dl), neoplasia.
11. SGPT, SGOT value greater than 2 times of the upper normal limit.
12. Insulin dependent diabetes mellitus or poorly controlled non-insulin dependent diabetes mellitus (AC sugar > 300 mg/dl).
13. Use of other anticoagulants, such as anti-coagulated agents or NSAIDsS.
14. History of alcohol and/or drug abuse.
15. Having participated in other investigational drug study within 3 months prior to study entry.
16. Pregnant or lactating women or women of childbearing potential whom are not practicing reliable birth control.
17. The patients who take methylxanthine-containing drinks or foods (coffee, black tea, cola, energy drink, etc.) more than 4 cups of coffee or it's equivalents.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2002-09; Primary Completion 2003-04 (Actual); Study Completion 2003-04

PRIMARY OUTCOMES:
Cumulated headache (intensity x frequency) over the first three days of treatment period

SECONDARY OUTCOMES:
Proportion of (1) subjects drop out due to drug related AE and (2) experiencing grade 3 or 4 drug related headache during day 5-14, day 15-21 (reduced dose), day 5-11 (regular dose), day 7, day 28; as well as (3) Number of acetaminophen tablets used.

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Taiwan Ltd.
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan